CLINICAL TRIAL: NCT05514925
Title: Peripheral Retinal Cryoapplication Versus Anti-VEGF Intravitreal Injection Before Vitrectomy for Complicated Proliferative Diabetic Retinopathy
Brief Title: Cryoapplication Versus Anti-VEGF Before Diabetic Vitrectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khairallah Moncef (Other)
Responsible Party: Sponsor-Investigator, Khairallah Moncef, Clinical Professor, University Hospital Fattouma Bourguiba
Organization: University Hospital Fattouma Bourguiba (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LR18SP09 N01; IORG0009738 N95 (Registry Identifier: Medicine Faculty of Monastir, Monastir University)
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Proliferative Diabetic Retinopathy; Vitreous Hemorrhage; Tractional Retinal Detachment
Keywords: Retinal cryoapplication; Anti-VEGF; Vitrectomy
MeSH Terms: conditions — Vitreous Hemorrhage | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative Anti-VEGF Intravitreal Injection (Active Comparator): Three to five days before vitrectomy, each participant received one intravitreal Bevacizumab injection (1.25 mg,0.05 ml).
  Interventions: Drug: Bevacizumab Injection [Avastin]
- Peripheral Retinal Cryoapplication (Experimental): Four to six weeks before vitrectomy, each participant underwent peripheral retinal cryoapplication.
  Interventions: Procedure: Peripheral Retinal Cryoapplication

INTERVENTIONS:
Drug: Bevacizumab Injection [Avastin] — Intravitreal injection of bevacizumab (1.25 mg, 0.05 ml) in the inferior temporal quadrant of the eye, 4 mm behind the limbus in phakic eyes, and 3.5 mm in pseudophakic eyes.
  Other Names: IVB
  Arms: Preoperative Anti-VEGF Intravitreal Injection
Procedure: Peripheral Retinal Cryoapplication — In the operating room under peribulbar anesthesia, four focal conjunctival incisions are made on each quadrant between the muscles insertions. The Tenon capsule is opened with scissors to expose the sclera. Four to six cryo-applications are made per quadrant, at the edge of muscle insertion and a line behind. The exposure time is 4 to 5 seconds. 7-0 resorbable sutures are then put on each quadrant to close the conjunctiva.
  Other Names: CRYO
  Arms: Peripheral Retinal Cryoapplication

SUMMARY:
Pars-plana vitrectomy (PPV) is the cornerstone of surgical treatment for eyes with complicated proliferative diabetic retinopathy. Anti-VEGF intravitreal injection before PPV has shown a good effect on surgical outcomes. However, many patients present with co-morbidities that contraindicate the usage of anti-VEGF in the pre-operative period. Thus, cryoapplication, an old therapeutic tool for proliferative diabetic retinopathy may be a good alternative. The investigators present herein a comparative study between peripheral retinal cryoapplication and anti-VEGF before vitrectomy for complicated proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
Pars-plana vitrectomy (PPV) is the cornerstone of surgical treatment of complicated proliferative diabetic retinopathy allowing the removal of vitreous opacity and releasing tractions from the retina. Surgical outcomes, however, are variable depending on a large array of pre, per, and post-operative conditions.

The preoperative anti-VEGF intravitreal injection has shown a good effect on surgical outcomes in patients with vitreous hemorrhage or tractional retinal detachment.

However, a great number of patients present with co-morbidities that contraindicate the usage of anti-VEGF in the pre-operative period.

Thus, an alternative to this adjunctive therapy is worth investigating. In another hand, cryoapplication, an old therapeutic tool for proliferative diabetic retinopathy had been used in patients with non-clear ocular media with vitreous hemorrhage.

The investigators present herein a comparative study between peripheral retinal cryoapplication and anti-VEGF before vitrectomy for complicated proliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Vitreous or retro-hyaloidal hemorrhage and/or tractional retinal detachment threatening or involving the macula
* No or less than 1000 impacts of preoperative retinal photocoagulation and/or iris rubeosis
* Only one eye per participant

Exclusion Criteria:

* Negative light perception
* Previous vitrectomy
* Contraindication to anti-VEGF therapy or retinal cryoapplication
* Associated rhegmatogenous retinal detachment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-11-21 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Total surgical time | at the end of the vitrectomy
  Duration of vitrectomy from the placement of the trocars until their removal
Intraoperative bleeding | at the end of the vitrectomy
  occurrence of intravitreal bleeding during vitrectomy

SECONDARY OUTCOMES:
Postoperative bleeding | one month after the vitrectomy
  occurrence of intravitreal bleeding after vitrectomy
Visual acuity | one month after the vitrectomy
  Best corrected logMAR visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Imen Ksiaa, Assoc. Prof., Principal Investigator — Fattouma Bourguiba University Hospital
Locations (1):
- Fattouma Bourguiba University Hospital - Ophthalmology Department, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang ZH, Liu HY, Hernandez-Da Mota SE, Romano MR, Falavarjani KG, Ahmadieh H, Xu X, Liu K. Vitrectomy with or without preoperative intravitreal bevacizumab for proliferative diabetic retinopathy: a meta-analysis of randomized controlled trials. Am J Ophthalmol. 2013 Jul;156(1):106-115.e2. doi: 10.1016/j.ajo.2013.02.008. PMID 23791371
- [Background] Arevalo JF, Lasave AF, Kozak I, Al Rashaed S, Al Kahtani E, Maia M, Farah ME, Cutolo C, Brito M, Osorio C, Navarro P, Wu L, Berrocal MH, Morales-Canton V, Serrano MA, Graue-Wiechers F, Sabrosa NA, Alezzandrini AA, Gallego-Pinazo R; Pan-American Collaborative Retina Study (PACORES) Group. Preoperative Bevacizumab for Tractional Retinal Detachment in Proliferative Diabetic Retinopathy: A Prospective Randomized Clinical Trial. Am J Ophthalmol. 2019 Nov;207:279-287. doi: 10.1016/j.ajo.2019.05.007. Epub 2019 May 13. PMID 31095954
- [Background] Lim AS, Ang BC. Cryoapplication in diabetic retinopathy. Int Ophthalmol. 1986 May;9(2-3):139-41. doi: 10.1007/BF00159842. PMID 3721714